CLINICAL TRIAL: NCT05958394
Title: Communication Training Around Sexual Health Topics for Parents of Youth With Autism Spectrum Disorder
Brief Title: Evaluation of Skillflix for Parents of Youth With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ashley Philliber (Other)
Collaborators: dfusion Inc (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Ashley Philliber, Managing Director, Philliber Research & Evaluation
Organization: Philliber Research & Evaluation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R43ES024563
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder (ASD); MicroSkills; Video training; Sexual and Reproductive Health; Parent Child Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): This arm will receive the intervention. This intervention is access to the SkillFlix for Parents Microskills video library, about 60 minute in duration. The library includes a curriculum covering skills such as seizing teachable moments, talking about identities, and using a conversation tone.
  Interventions: Behavioral: SkillFlix for Parents
- Control (No Intervention): During the intervention period arm 2 will receive written conversation guides for the assigned conversations. This arm will receive the intervention upon completion of follow-up study activities.

INTERVENTIONS:
Behavioral: SkillFlix for Parents — A Microskills video training library on communication skills for talking to youth about relationships and sexual health topics.
  Arms: Treatment

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of using a Microskills video training library for training parents of adolescents with ASD in talking with their teens about relationships and sexual health topics.

The main questions it aims to answer are:

* Does using SkillTalk increase parents' skills in communicating with their teens about relationships and sexual health?
* Does using SkillTalk increase the frequency of conversations about relationships and sexual health?
* Does using SkillTalk increase parents' confidence in their ability to communicate with their teens about relationships and sexual health?
* Does using SkillTalk improve teen knowledge, attitudes, and behavior around sexual health and relationships?

Participants will be asked to:

* Take a survey at the beginning of the study, the end of the study, and at 3-month follow up
* Record a short conversation between the parent and teen dyad about a sexual health topic at the beginning of the study, at the end of the study, and at 3-month follow up.
* Watch a minimum of 85% of the 60 minutes of video assigned
* Complete a conversation log at the end of each week during the study period, and once a month during the 3-month follow-up period.

DETAILED DESCRIPTION:
The proposed project will establish the efficacy of using the SkillFlix for Parents online video library to improve the sexual health communication skills of parents of teens with autism spectrum disorder. A randomized controlled trial is being conducted to assess the impact of the resource on parent skill demonstration and confidence, conversation frequency, and teen knowledge, attitudes, and behaviors. Participants will be parent and youth dyads, including parents over 18 years old and youth aged 13-17 with ASD, reciprocal communication skills, receptive language skills, who are in mainstream classrooms for at least one class during the school day.

Participants are primarily being recruited with assistance from agencies/organizations that serve those with ASD, community and professional advisory board members, and other community networks. It is also likely that participants will refer other parents of youth on the spectrum for participation.

The study design will be a randomized controlled trial of dyads with pre- and post-assessment, and a 3-month follow-up assessment (6 months after start of study), each including a survey and audio recording. After completing the baseline activities, half (50) of the dyads will be randomly assigned to the SkillTalk ASD intervention group which will receive access to the SkillTalk ASD web site and the study mobile app. The control group will receive written materials with similar content. For baseline parents will take a survey, audio record a conversation based on a written conversation guide and upload it for analysis. Youth will take a survey. Intervention participants will have access to SkillTalk ASD for 3 months. During the three-month period, parent and youth participants will be asked to complete a bi-weekly conversation log. At the conclusion of the three-month period, they will participate in an immediate post-test which will again include a survey, audio record a conversation based on a written conversation guide and upload it for analysis. Youth will take an immediate post-test survey. During the three-month follow-up period, parents and youths will be asked to complete a biweekly conversation log. Three months after the conclusion of the access period parents will take a survey, audio record a conversation based on a written conversation guide and upload it for analysis. Youth will take a survey. At the conclusion of the 6-month period the control group participants will be provided with access to the SkillFlix ASD materials.

ELIGIBILITY:
Inclusion Criteria:

* Eligible dyads will:

  * Have a parent of youth aged 13-17 with diagnosed ASD.
  * Have a child aged 13-17 with ASD. The child must:

    * have reciprocal communication skills and receptive communication skills
    * be in mainstream classrooms for a minimum of one class during the school day
  * Have access to a computer/mobile device connected to the internet.

Exclusion Criteria:

* There will be no exclusionary criteria based on gender or race/ethnicity, however during recruitment and enrollment staff will try to ensure that the race/ethnicity demographics reflect those of the U.S. more generally, with a 10% oversampling for Black and Latinx participants, and the gender ratio is balanced. Parent participants will not be screened for or included/excluded on the basis of having ASD themselves.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Demonstrated Skill score in communicating with their teens about sexual health | 3 months
  Based on a rubric created for this study of the demonstrable skills for the given recorded conversation topic. The points earned on the rubric are summed to create a total score. The scale ranges from 0 to 20 with a higher score indicating higher skill usage.

SECONDARY OUTCOMES:
Parent reported frequency of discussions with their teens about sexual health and relationships over the course of the last 3 months. | 3 months
  Frequency will be broken down by topic into Relationships, Puberty, Public/Private, Sexual Health, Personal Safety, STIs.
Parent Conversation Quality Score | 3 months
  Based on a scale created for this study, the Conversation Quality Score is comprised of a series of conversation log questions about teen engagement and perceived effectiveness of the conversation. The scores from the question are summed to create a total score. The score range is 3 to 15 with higher scores indicating a high quality of conversation.
Parent confidence in their ability to use skills in communication with their teen about sexual health and relationships. | 3 months
  Based on a scale created for the study, the score is comprised of a series of questions about ability to discuss safer sex topics, use a conversational tone, practice active listening, answer questions, and navigate teen readiness. The scores from the question are summed to create a total score. The score range is 5 to 25, with higher scores indicating more confidence in ability.
Parent confidence in teens ability to use Making Connections skills. | 3 months
  Based on a scale created for the study, the score is comprised of a series of questions about ability to use effective communication techniques with trusted adults, have challenging conversations with adults, seize askable moments, and establish boundaries. The scores from the question are summed to create a total score. The score range is 4 to 20, with higher scores indicating more confidence in ability.
Teen reported frequency of discussions with their teens about sexual health and relationships over the course of the last 3 months. | 3 months
  Frequency will be broken down by topic into Relationships, Puberty, Public/Private, Sexual Health, Personal Safety, STIs.
Youth Conversation Quality Score. | 3 months
  Based on a simple 5 point rating system. The score range is 1-5, with higher scores indicating higher quality conversation.
Teen confidence in their ability to use Making Connections skills. | 3 months
  Based on a scale created for the study, the score is comprised of a series of questions about ability to use effective communication techniques with trusted adults, have challenging conversations with adults, seize askable moments, and establish boundaries. The scores from the question are summed to create a total score. The score range is 4 to 20, with higher scores indicating more confidence in ability.
Family Sex Communication Quotient Score | 3 months
  Based on a scale developed as a diagnostic tool to measure a general family orientation to discussion about sex between parents and children (Warren & Neer, 1982, 1983). The scores from the question are summed to create a total score. The score range is 18 to 90, with higher scores indicating high communication orientation.
Teen's Sexual Health Knowledge | 3 months
  Based on a scale created for this study, this score is comprised of a series of questions about the sexual health topics discussed in the recorded conversations. The scores from the question are summed to create a total score. The scale ranges from 0 to 5 with a higher score indicating greater knowledge.
Teen's sexual health attitudes | 3 months
  Based on a scale created for this study, this score is comprised of a series of questions about teens comfort regarding sexual health topics. The scores from the question are summed to create a total score. The scale ranges from 2 to 10 with a higher score indicating greater comfort.
Teen's sexual health behaviors | 3 months
  A series of questions about teens sexual health behaviors such as condom use, STI testing, and contraceptive use.

IPD SHARING:
Plan to Share IPD: No